CLINICAL TRIAL: NCT01394575
Title: Phase 2 Study of Whole Breast Irradiation With Inversely Intensity Modulated Radiotherapy and Simultaneously Integrated Boost for Early Stage Breast Cancer Patients
Brief Title: Whole Breast Irradiation With Intensity Modulated Radiotherapy and Simultaneously Integrated Boost for Early Stage Breast Cancer Patients
Acronym: IMRT-SIB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: The Department of Radiation Oncology, Fudan University Cancer Hospital, Fudan University Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-RT-001
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiotherapy; simultaneous integrated boost; tumor bed; IMRT
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT-SIB (Experimental)
  Interventions: Radiation: IMRT with an simultaneous integrated boost

INTERVENTIONS:
Radiation: IMRT with an simultaneous integrated boost — IMRT in 25 fractions delivering 45Gy to the whole breast and 60Gy to the tumor bed

SUMMARY:
This is a phase II study. In patients with node-negative invasive breast cancer or carcinoma in situ treated by breast conserving surgery, postoperative whole breast irradiation with inversely intensity modulated radiotherapy and a simultaneous integrated boost is technically feasible. The aim of this study is to evaluate the radiation toxicity, cosmetic outcome and local control rate in a single center

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance score﹤2
* All patients aged >18 years and < 70 years after breast conserving surgery.
* On histological examination, the tumor must be DCIS or invasive adenocarcinoma of the breast.
* Negative nodal status determined by sentinel node biopsy, or axillary dissection. Axillary staging is not required for patients with DCIS
* No evidence of distant metastasis
* Gross disease may be unifocal or multifocal with pathologic (invasive and/or DCIS) tumor size excised with negative margins（>2mm）
* Surgical treatment of the breast must have been lumpectomy. Re-excision of surgical margins is permitted.
* The patient must consent to be in the study and must have signed an approved consent form.

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance score≧2
* Presence of extensive intraductal component (ductal carcinoma in situ occupying > 25% of the primary invasive tumour and present adjacent to the primary tumour).Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
* Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant of separated.
* Metastatic disease (M1)
* Pregnancy or lactating
* Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation.
* Psychiatric or addictive disorders that preclude obtaining informed consent or adherence to protocol.
* Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
* Prior breast or thoracic RT for any condition.
* Previous or concomitant malignancies except non-melanoma skin cancer, carcinoma in situ of the cervix, and invasive carcinoma of the colon, thyroid, cervix, or endometrium treated five years prior to study entry.
* Synchronous chemotherapy or target therapy is not permitted.
* Refusal of the patients to be included in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Radiation toxicity | first analysis will occur 2 year after accrual of all patients
Cosmetic outcome | first analysis will occur 2 year after accrual of all patients

SECONDARY OUTCOMES:
Time to ipsilateral breast recurrence | first analysis will occur 5 year after accrual of all patients
Local recurrence rate | first analysis will occur 5 year after accrual of all patients
Disease free survival | first analysis will occur 5 year after accrual of all patients
Overall survival | first analysis will occur 5 year after accrual of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, MD, Principal Investigator — The Department of Radiation Oncology, Fudan University Cancer Hospital
Locations (1):
- The Department of Radiation Oncology,Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China